CLINICAL TRIAL: NCT03493152
Title: Expanded Access to Everolimus, for an Individual Patient With GIST (Gastrointestinal Stromal Tumors)(CTMS#18-0019)
Status: No longer available | Type: Expanded Access
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS# 18-0019; HSC20180169T (Other: UT Health San Antonio)
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Everolimus

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Everolimus — mTOR inhibitor
  Other Names: Zortress, Afinitor, and Afinitor Disperz

SUMMARY:
Single patient treatment with everolimus.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult